CLINICAL TRIAL: NCT04217850
Title: Efficacy of microRNA Testing for Identification of Personalized Weight Management Strategy in Obese and Overweight Individuals.
Brief Title: microRNA Testing for Identification of Personalized Weight Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: North Dakota State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EN20014
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Overweight and Obesity; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 500 kcal Energy Deficit (Experimental): The goal of the nutrition and exercise intervention will be to induce an energy deficit of approximately 500 kcals/day over the 12-week period in order to induce an approximate 5% weight loss in all participants.
  Interventions: Other: 250 kcal Dietary Energy Restriction; Other: Aerobic Exercise

INTERVENTIONS:
Other: 250 kcal Dietary Energy Restriction — The nutrition intervention will be individualized and implemented as a free-living energy-restricted eating plan where energy intake will be based on a mild restriction (approx. 250 kcal/day).
Other: Aerobic Exercise — Supervised aerobic exercise will be combined with the energy restriction. Individuals will perform aerobic exercise (treadmill, cycle, or rower or combination) 4-5 days per week for 12 weeks. At each session they will expend 250 or more calories to further meet or exceed the 500 kcal energy deficit.

SUMMARY:
Certain blood markers are related to one's ability to successfully lose weight by diet and exercise. Currently, the laboratory tests used to measure these blood markers are expensive and time-consuming. Recently, the Electrical and Computer Engineering Department, at NDSU, invented a device that may be able to measure these blood markers much more quickly and affordably. This study is designed participate, to compare our new device to previous methods. If the new sensor is successful, it will be used as diagnostic tool to personalize weight loss strategies.

DETAILED DESCRIPTION:
Obesity is increasing exponentially in the United States (US), and over 160 million Americans are either overweight or obese. A combined diet and exercise program is the most cost-effective alternative for weight management, but there is a considerable inter-individual variability in losing weight via this method, which leaves many individuals frustrated and unable to adhere to programs throughout the lifespan. Therefore, the inability to identify the individuals who will likely succeed with diet and exercise for weight management is a critical roadblock to treating obesity. Recent studies have shown that significant variability in weight loss response to diet and exercise could be attributed in part to individual epigenetic makeup. One potential approach for monitoring the epigenetic response during weight-loss interventions is small non-coding circulating RNAs, called microRNAs (miRNAs or miRs), in the circulating blood. Studies have shown that miR-140 and 935 could be used as blood biomarkers to identify individuals who will succeed in managing their weight through diet and exercise. Moreover, during a short diet and exercise intervention, fluctuations of expression levels of biomarker miRNAs pre- and post-intervention have produced unique signature changes only in the individuals who continued the intervention for an extended period of time and attained a healthy body weight. Thus, if implemented early in a medical weight loss program it could allow for the patient to have a focused individualized treatment.

A major barrier that prevents the use of miRNAs in weight loss interventions is the inability of accurately quantifying miR-140 and 935 levels in blood samples. To minimize the miRNA contamination from red-blood cell lysis, miRNA analysis must be performed within 30 minutes of blood draw. Current miRNA detection and quantification technologies take hours/days to quantify miRNAs, require bulky equipment, and are expensive. In addition, current miRNA detection methods do not have sufficient sensitivity, detection span and specificity for clinical sample analysis. To address this need, PI. Nawarathna has recently developed a highly sensitive disposable miRNA sensor that can quantify miRNAs in point-of-care settings within 15 minutes with an assay cost of $50 per test. However, the effectiveness of the developed miRNA sensor to accurately quantify the variations of target miRNA levels (miR-140 and 935) pre- and post-diet and exercise intervention is unknown.

The objective of the proposed work is to investigate the efficacy of this miRNA sensor as a potential diagnostic device in weight management. If successful, the impact of proposed the research is two-fold: first, development of a point-of-care diagnostic device (miRNA sensor) for providing a personalized strategy for weight management (diet and exercise or bariatric surgery) and second, ability to immediately expand miRNA detection to measure other factors that can impact overall well-being (e.g.: mental and emotional health, stress, and fatigue) and diseases (e.g.: cancer, cardiovascular diseases, and others). The objective of the proposed research will be achieved through following this specific aim:

Aim: To investigate if the miRNA sensor is capable of identifying individuals who will consistently lose weight with energy restricted diet and exercise intervention.

The proposed research will develop a pilot study with overweight individuals as participants. Subjects will participate in the diet and exercise intervention for 12 weeks and miRNA analysis will be performed at 3 time points during the intervention (pre-mid-post). We will then investigate the effectiveness of the sensor.

The miRNA sensor technology, once fully developed, will be similar to a finger prick glucose monitor. Once commercially available, miRNA sensors can be purchased and used for diagnostic applications in clinics or self-testing at home or remote and rural area clinics and hospitals. Therefore, the outcomes will fundamentally advance how the individualized weight management method is selected. For this reason, this research has a positive translational impact on human health.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* body mass index 25-34.9
* able to do physical activity and exercise

Exclusion Criteria:

* currently participating in a structured diet or excise program,
* pregnant,
* currently use any nicotine product
* diagnosed neuromuscular disease
* diabetes,
* uncontrolled high blood pressure,
* diagnosed cancer,
* previously had a heart attack or other chronic heart related conditions that are not controlled with medicine
* difficulty moving without assistive devices or walking one-quarter mile
* are taking medications that influence muscle size (testosterone, growth hormone, etc.),
* have had bariatric surgery
* have a body mass greater than 350lbs,
* fear blood, blood draws, or needles
* adverse reaction to a blood draw in the past.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
micro RNA 140 | Change across weeks 0, 6, 13
  Venous blood concentrations (M) of micro RNA 140 will be measured using our sensor.
micro RNA 935 | Change across weeks 0, 6, 13
  Venous blood concentrations (M) of micro RNA 935 will be measured using our sensor.
Body Composition | Change across weeks 0, 6, 13
  Change in body composition (% fat) derived from dual x-ray absorptiometry
Lean body mass | Change across weeks 0, 6, 13
  Change in lean body mass (kg) derived from dual x-ray absorptiometry
Fat mass | Change across weeks 0, 6, 13
  Change in fat mass (kg) derived from dual x-ray absorptiometry
Body mass | Change across weeks 0, 6, 13
  Change in body mass (kg) derived from scale

SECONDARY OUTCOMES:
High-density lipoprotein | Change across weeks 0, 6, 13
  Change in high density lipoprotein (mg/dL) from Piccolo Xpress Blood Chemistry Analyzer
Total cholesterol | Change across weeks 0, 6, 13
  Change in total cholesterol (mg/dL) from Piccolo Xpress Blood Chemistry Analyzer
Triglycerides | Change across weeks 0, 6, 13
  Change in triglycerides (mg/dL) from Piccolo Xpress Blood Chemistry Analyzer
Low-density lipoprotein (calculated) | Change across weeks 0, 6, 13
  Change in low-density lipoprotein (mg/dL) from Piccolo Xpress Blood Chemistry Analyzer
Very low-density lipoprotein (calculated) | Change across weeks 0, 6, 13
  Change in very low-density lipoprotein (mg/dL) from Piccolo Xpress Blood Chemistry Analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States